CLINICAL TRIAL: NCT04695938
Title: Craniofacial Imaging With 3D MRI: an Alternative to Ionising Radiation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cambridge (Other)
Collaborators: Great Ormond Street Hospital for Children NHS Foundation Trust (Other); Oxford University Hospitals NHS Trust (Other); Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr Karen A Eley, Clinical Lecturer in Radiology, University of Cambridge
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18/WA/0155
Record Dates: First submitted 2020-02-07; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Craniosynostoses; Synostosis; Skull Deformity
Keywords: Image Reconstruction; Medical Imaging; Magnetic Resonance Imaging; Imaging, Three-Dimensional
MeSH Terms: conditions — Craniosynostoses; Synostosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI (Other): MRI examination
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — MRI examination with Black Bone, and ultrashort/zero echo time MRI techniques

SUMMARY:
Craniosynostosis is a condition where infants are born with or subsequently develop an abnormally shaped skull. The skull develops from plates of bone separated from each other by growth lines (sutures). Craniosynostosis refers to early fusion of one or more of these sutures.

Whilst in many cases the abnormal head shape provides doctors with the underlying diagnosis, it is necessary to confirm this using imaging. A CT scan involves using multiple x-rays to build a picture of the part of the body being examined. X-rays are associated with potential long term harm, particularly in young children who have longer to incur those risks. MRI uses magnets and radiowaves to create images of the body, and therefore a radiation-free method of imaging.

The investigators have previously shown in a pilot group that a specific MRI technique ("Black Bone") can distinguish between normal and prematurely fused cranial sutures, and that the images can be reconstructed in 3D in the same way as CT.

The investigators now need to confirm the findings in a larger patient group, and develop automated methods of creating 3D images of the bone.

Children in whom there is clinical suspicion of craniosynostosis will be recruited for MRI examination. In children who are already undergoing MRI examination of the head (for any indication), the investigators will add on bone specific sequences.

There are no known long term risks associated with MRI, and no contrast medium is required. Anonymised MRI data will be used to further develop our 3D techniques.

ELIGIBILITY:
Inclusion Criteria:

* Children in whom craniosynostosis is clinically suspected

Exclusion Criteria:

* Children with contraindications to MRI examination
* Children who require sedation/anaesthesia solely for the purpose of research MRI

Ages: 0 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2020-11-27 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of craniosynostosis | Average one week for diagnosis of individual participants. End of study (2 years) for cohort analysis.
  Accuracy of diagnosis on MRI of craniosynostosis
3D reconstruction of craniofacial MRI | Preliminary 3D outputs within 2 weeks of participation per patient, and by end of study for automated segmentation algorithms(2 years)
  Automated segmentation of craniofacial MRI

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cambridge, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided